CLINICAL TRIAL: NCT07186101
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Active-Controlled Study of LY4268989 (MORF-057) Co-Administered With Mirikizumab in Adults With Moderately to Severely Active Ulcerative Colitis
Brief Title: LY4268989 (MORF-057) Co-Administered With Mirikizumab in Adults With Moderately to Severely Active Ulcerative Colitis:
Acronym: TOPAZ-UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27704; J6E-MC-KWAN (Other: Eli Lilly and Company); MORF-057 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY4268989 + Mirikizumab (Experimental): LY4268989 administered orally (PO) + Mirikizumab administered intravenously (IV), then subcutaneously (SC). Responders will be re-randomized for Study Period 2.
  Interventions: Drug: LY4268989; Drug: Mirikizumab
- Mirikizumab + LY4268989 Placebo (Experimental): Mirikizumab administered IV, then SC + LY4268989 placebo administered PO. Responders and Non-responders will re-randomized for Study Period 2.
  Interventions: Drug: Mirikizumab; Drug: LY4268989 Placebo

INTERVENTIONS:
Drug: LY4268989 — Administered PO
  Other Names: MORF-057
  Arms: LY4268989 + Mirikizumab
Drug: Mirikizumab — Administered IV then SC
  Other Names: LY3074828
Drug: LY4268989 Placebo — Administered PO
  Arms: Mirikizumab + LY4268989 Placebo

SUMMARY:
The main purpose of the study is to evaluate the effectiveness and safety of LY4268989 when given with mirikizumab compared to mirikizumab alone in adult participants with moderately to severely active ulcerative colitis (UC).

Study participation will last approximately 118 weeks, including 104 weeks of treatment and may include up to 21 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have had an established diagnosis of ulcerative colitis (UC) of ≥3 months in before baseline, which includes endoscopic evidence of UC and a histopathology report that supports a diagnosis of UC
* Have moderately to severely active UC as defined by a Modified Mayo Score (mMS) of 5 to 9 with an Endoscopic Score (ES) ≥2 confirmed by central reader and rectal bleeding (RB) ≥1, with endoscopy performed within 21 days before baseline
* Participants with greater than 8 years of UC symptoms have documented evidence of having had a surveillance colonoscopy within 1 year, or according to local country or regional medical guidelines, to evaluate for polyps, dysplasia, or malignancy, prior to randomization
* Are up-to-date on colorectal cancer surveillance per local society guidelines
* Have an inadequate response to, loss of response to, or intolerance to at least 1 of the medications:
* Conventional-failed participants: Participants who have had an inadequate response to or a loss of response to or are intolerant to at least 1 of the following medications: corticosteroids or immunomodulators (Does not apply to US)

NOTE: After the interim analysis, participants with inadequate response, loss of response, or intolerance to conventional UC therapy without prior exposure to biologics may be enrolled if deemed appropriate (Applies to the US)

* Advanced therapy-failed participants: Participants who have an inadequate response to or a loss of response to, or are intolerant to advanced therapy for UC, defined as:

  * a biologic or biosimilar medication such as anti-tumor necrosis factor (anti-TNF) antibodies or anti-interleukin antibodies (IL-12/23, or IL-23p19), except for

    * mirikizumab.
  * Janus kinase inhibitors (JAK) such as filgotinib, tofacitinib, or upadacitinib
  * sphingosine 1-phosphate receptor 1 inhibitors (S1PR) such as etrasimod or ozanimod

Exclusion Criteria:

* Have a current diagnosis of

  * Crohn's disease
  * Inflammatory Bowel Disease (IBD) unclassified (formerly known as indeterminate colitis), or
  * primary sclerosing cholangitis
* Have had or will need bowel resection or intestinal or intra-abdominal surgery
* Have evidence of toxic megacolon, intra-abdominal abscess, or stricture or stenosis within small bowel or colon that cannot be traversed by a colonoscope or that are symptomatic
* Have any adenomatous polyp occurring in areas of the colon not involved by colitis, that has not been removed

Note: If such an adenomatous polyp has been completely removed and shows only low-grade dysplasia, this criterion would no longer apply

* Have a current or recent acute, active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve Clinical Remission with Modified Mayo Score (mMS) | Week 12
  The mMS is a composite sore reported by participants and physician and is comprised of the following 3 subscores: Stool Frequency (SF); Rectal Bleeding (RB), and Endoscopic Subscore (ES).
  Clinical remission (mMS) is defined as:
  * SF subscore = 0 or 1 and no greater than baseline
  * RB subscore = 0
  * Centrally read ES = 0 or 1; score of 1 modified to exclude friability

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve Clinical Response with Modified Mayo Score (mMS) | Week 12
Percentage of Participants Who Achieve Endoscopic Improvement | Week 12
Percentage of Participants Who Achieve Symptomatic Remission | Week 12
Percentage of Participants Who Achieve Clinical Remission with mMS | Week 24
Percentage of Participants Who Achieve Clinical Response with mMS | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (149):
- United States (40):
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - Clinnova Research - Anaheim, Anaheim, California
  - Om Research LLC, Lancaster, California
  - Biopharma Informatic, LLC, Los Angeles, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - NeoClinical Research, Hialeah, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Clinical Research of Osceola, Kissimmee, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Alliance Medical Research, Lighthouse PT, Florida
  - Atlantic Medical Research, Margate, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Center for Gastrointestinal Health - Fairview Heights, Belleville, Illinois
  - Midtown Gastroenterology and Liver Disease, Des Plaines, Illinois
  - GI Alliance - Glenview, Glenview, Illinois
  - Gi Alliance - Gurnee, Gurnee, Illinois
  - Gastroenterology Health Partners, New Albany, Indiana
  - Gastroenterology Health Partners, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Clinton Township, Michigan
  - GI Associates - GIA and Endoscopy Center - Flowood, Flowood, Mississippi
  - Columbia University Irving Medical Center, New York, New York
  - Digestive Disease Medicine of Central New York, Utica, New York
  - Gastroenterology & Hepatology Specialists, Canton, Ohio
  - Dayton Gastroenterology, LLC, Dayton, Ohio
  - University Gastroenterology - Providence - West River Street, Providence, Rhode Island
  - Gastroenterology Associates, P.A. of Greenville, Greenville, South Carolina
  - Gastro One - Walnut Run Road, Cordova, Tennessee
  - Texas Digestive Disease Consultants - Cedar Park, Cedar Park, Texas
  - GI Alliance - Dallas - Gaston Avenue, Dallas, Texas
  - GI Alliance - Fort Worth, Fort Worth, Texas
  - GI Alliance - Garland, Garland, Texas
  - GI Alliance - Lubbock, Lubbock, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - GI Alliance-Webster, Webster, Texas
  - Care Access - Ogden, Ogden, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
  - GI Alliance - Richmond, Richmond, Virginia
  - Washington Gastroenterology - Bellevue, Bellevue, Washington
- Austria (2):
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Brazil (13):
  - Chronos Pesquisa Clínica, Brasília
  - CAEP - Synvia Labs, Campinas
  - Fundação Universidade de Caxias do Sul (FUCS), Caxias do Sul
  - Centro Digestivo de Curitiba, Curitiba
  - Galileo Medical Research, Juiz de Fora
  - NewData Clinical Research - Maceió, Maceió
  - Hospital Ernesto Dornelles, Porto Alegre
  - Centro Internacional de Pesquisa Clínica (CIPES), São José dos Campos
  - CPQuali Pesquisa Clínica, São Paulo
  - Solare Trials, São Paulo
  - Hospital Santa Catarina - Paulista, São Paulo
  - Clínica Hepatogastro JK, São Paulo
  - Universidade Federal Do Piaui - Campos Universitario, Teresina
- Canada (5):
  - Charlton Digestive Disease Centre, Hamilton
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London
  - London Digestive Disease Institute, London
  - West GTA Research Inc., Mississauga
  - C.I.C. Mauricie inc., Trois-Rivières
- China (12):
  - Changzhou Second People's Hospital, Changzhou
  - Chongqing General Hospital, Chongqing
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Afilliated Hospital of Hebei Medical University, Shijiazhuang
  - Taian City Central Hospital, Taian
  - Wuhan Union Hospital, Wuhan
  - Wuxi People's Hospital, Wuxi
- Denmark (4):
  - Aalborg Universitetshospital, Syd, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Herlev and Gentofte Hospital, Copenhagen
  - Odense Universitetshospital, Odense
- Germany (4):
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Studienzentrum MVZ Dachau, Dachau
  - Universitätsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Ulm, Ulm
- Hungary (7):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannónia Magánorvosi Centrum, Budapest
  - Clinexpert Gyöngyös, Gyöngyös
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
  - Jávorszky Ödön Kórház, Vác
- India (8):
  - Sardar Vallabhbhai Patel Institute of Medical Sciences and Research, Ahmedabad
  - Rajiv Gandhi Government General Hospital, Chennai
  - Ashwin Hospital, Coimbatore
  - Sushruta Multispeciality Hospital & Research Centre, Hubli
  - Mahavir Hospital & Research Centre - Hyderabad, Hyderabad
  - All India Institute of Medical Sciences, New Delhi
  - Medipoint Hospitals Pvt. Ltd., Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
- Italy (5):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Humanitas, Rozzano
- Japan (6):
  - Fukuoka University Hospital, Fukuoka
  - Gokeikai Ofuna Chuo Hospital, Kamakura
  - Tsujinaka Hospital - Kashiwanoha, Kashiwa
  - National Hospital Organization Osaka National Hospital, Osaka
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
- Mexico (12):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Boca Clinical Trials Mexico S.C., Guadajalara
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - Centro de Investigación y Gastroenterología - S.C., Mexico City
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Servicios de Oncología Médica Integral - Monterrey, San Pedro Garza García
  - Scientia Investigacion Clinica S.C., Tijuana
  - Clinical Research Institute S.C., Tlalnepantla
  - Medimanage Research, Tlalpan
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (2):
  - Radboudumc, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- Poland (9):
  - Gyncentrum sp. z o.o. NZOZ Holsamed - oddział Libero, Katowice
  - IRMED, Piotrkow Trybunalski
  - Pratia Poznań, Poznan
  - Uniwersyteckie Centrum Stomatologii i Medycyny Specjalistycznej, Poznan
  - Twoja Przychodnia SCM, Szczecin
  - Sonomed Sp. z o. o., Szczecin
  - WSD MEDI, Warsaw
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - ETG Zamość, Zamość
- Romania (6):
  - Spitalul de Oncologie Monza, Bucharest
  - Delta Health Care, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Constanta County Emergency Clinical Hospital Sf.Ap.Andrei, Constanța
  - Spital Judetean de Urgenta, Satu Mare
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Spain (5):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital de Cabueñes, Gijón
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Eskisehir Osmangazi University, Eskişehir
  - Mustafa Kemal Universitesi, Hatay
  - Kocaeli University Medical Faculty Hospital, İzmit
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi, Malatya
  - Mersin University, Mersin
  - Dicle Üniversitesi, Sur

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: LY4268989 (MORF-057) Co-Administered With Mirikizumab in Adults With Moderately to Severely Active Ulcerative Colitis: (TOPAZ-UC) — https://trials.lilly.com/en-US/trial/655156